CLINICAL TRIAL: NCT04841356
Title: Swelling Management After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Joint Replacement (Other); medi (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1722208-1
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Total Knee Arthroplasty
Keywords: swelling; compression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICG (Experimental): Immediate Compression Garment
  Interventions: Procedure: Immediate Compression Garment

INTERVENTIONS:
Procedure: Immediate Compression Garment — Immediately following surgery, in the operating room, the compression garment will be donned on the surgical limb. The garment is set to the following pressures to facilitate gradient compression: 40mm Hg (lower leg), 30mm Hg (knee), 20 mm Hg (thigh) utilizing a standardized garment tensioning tool. Subjects will wear the garment during all waking hours (target wear time of 12 hours daily) for the first 3 weeks after surgery. Additionally, subjects will be instructed to perform a therapeutic exercise program designed to manage swelling by targeting major lower extremity musculature (gastrocnemius, soleus, quadriceps, hamstrings, and gluteal musculature) and promoting venous and lymphatic return. These exercises will be performed five times daily during the first three weeks after surgery.
  Subjects will receive standard of care rehabilitation following surgery as directed and coordinated by the surgeon and participant. This rehabilitation is not part of this research study.
  Other Names: compression

SUMMARY:
The purpose of this feasibility study is to estimate the initial efficacy and feasibility of an inelastic compression garment donned immediately after TKA on peak swelling in 14 subjects.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is the most commonly performed surgical procedure in older adults and is expected to increase five-fold by 2040 to 3.5 million TKAs annually. Although TKA is effective at reducing pain and improving self-reported quality of life, postoperative knee swelling after TKA is profound with the average level of swelling peaking at a 35% increase in the first 6-8 days after surgery and persisting months after surgery. Postoperative swelling is associated with a 60% decrease in quadriceps strength in the first month after surgery leading to decreases in functional performance of up to 90%. Patients can exhibit chronic strength deficits on the order of 28-42% based on comparisons with age-matched controls years after surgery. Quadriceps weakness results in long-term decreases in gait speed, balance, stair-climbing ability, chair rise ability, increased risk for falls and disability later in life. Additionally, postoperative knee swelling has also been associated with increased pain, decreased range of motion (ROM) and post-surgical complications such as deep venous thrombosis (DVT) and infection. Traditional postoperative interventions such as elastic compression stockings (e.g., thromboembolism-deterrent (TED) hose) have demonstrated minimal effectiveness in reducing swelling after TKA. We have demonstrated in a preliminary study (N=16) that an inelastic, adjustable compression garment, commonly utilized to manage patients with chronic lymphedema, can decrease postoperative cumulative swelling by 50% in the early postoperative period. With this data, the garment was not applied until postoperative day 4 and thus it had minimal effect on the peak swelling noted after surgery. Peak swelling, not cumulative, is associated with strength and function after TKA. Therefore, this feasibility study aims to mitigate peak swelling by donning the compression garment immediately after surgery in the operating room. It also seeks to assess the feasibility of the intervention from the subjects' perspective.

Specific Aim 1:

Estimate the effect of immediate compression garment (ICG) on the primary outcome of swelling at 4 days and 1, 2, 3, and 6 weeks postoperative.

Hypothesis: The ICG group will have less swelling at 4 days and 1, 2, 3, and 6 weeks postoperative compared to historical controls.

Specific Aim 2:

Determine the participant feasibility of ICG by assessing 1) satisfaction and 2) adherence.

Hypothesis 3.1: Study participants will indicate acceptability of compression garment wear with a median score of at least 4/5 ("somewhat satisfied") on a 5-point Likert scale satisfaction survey.

Hypothesis 3.2: An 80% adherence rate will be observed for compression garment wear as assessed by a patient log.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo a primary, unilateral total knee arthroplasty secondary to end-stage osteoarthritis

Exclusion Criteria:

* Discharge to location other than home after surgery
* History of heart failure, lymphatic insufficiency, hepatic disease, pre-existing pitting edema, varicose vein ligation or any other condition associated with lower extremity swelling
* Unstable orthopedic conditions (besides OA/TKA) that limit function
* Other neurological, vascular, or cardiac problems that limit function or cause chronic lower extremity swelling
* No caregiver or inability to touch toes which can affect the ability to don/doff the compression garment
* Current smoker or history of substance abuse
* Surgical complication necessitating an altered course of rehabilitation
* Uncontrolled diabetes (hemoglobin A1c level >8.0)
* Body mass index >40 kg/m2

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Change in total limb swelling from baseline to day 4 and weeks 1, 2, 3, and 6 postoperative | preoperatively, day 4 and weeks 1, 2, 3, and 6 postoperatively
  Assesses swelling in the lower extremity using single frequency bioelectrical impedance.

SECONDARY OUTCOMES:
Adherence to the intervention as measured by self-report logs | week 3 postoperatively
  Adherence will be calculated from 0-100% by taking the total number of days the garment was worn for 12+ hours divided by the total number of possible days. Informs feasibility of intervention.
Subject satisfaction as measured by a 5-point Likert scale ranging from "very unsatisfied" to "very satisfied" | week 3 postoperatively
  Assesses the satisfaction of subjects with the intervention using a 5-point Likert scale ranging from "very unsatisfied" to "very satisfied". Informs feasibility of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Jennings, MD, Principal Investigator — Colorado Joint Replacement
Locations (1):
- Colorado Joint Replacement, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh JA, Yu S, Chen L, Cleveland JD. Rates of Total Joint Replacement in the United States: Future Projections to 2020-2040 Using the National Inpatient Sample. J Rheumatol. 2019 Sep;46(9):1134-1140. doi: 10.3899/jrheum.170990. Epub 2019 Apr 15. PMID 30988126
- [Background] Loyd BJ, Kittelson AJ, Forster J, Stackhouse S, Stevens-Lapsley J. Development of a reference chart to monitor postoperative swelling following total knee arthroplasty. Disabil Rehabil. 2020 Jun;42(12):1767-1774. doi: 10.1080/09638288.2018.1534005. Epub 2019 Jan 22. PMID 30668214
- [Background] Bade MJ, Kohrt WM, Stevens-Lapsley JE. Outcomes before and after total knee arthroplasty compared to healthy adults. J Orthop Sports Phys Ther. 2010 Sep;40(9):559-67. doi: 10.2519/jospt.2010.3317. PMID 20710093
- [Background] Loyd BJ, Stackhouse S, Dayton M, Hogan C, Bade M, Stevens-Lapsley J. The relationship between lower extremity swelling, quadriceps strength, and functional performance following total knee arthroplasty. Knee. 2019 Mar;26(2):382-391. doi: 10.1016/j.knee.2019.01.012. Epub 2019 Feb 14. PMID 30772186
- [Background] Huang CH, Cheng CK, Lee YT, Lee KS. Muscle strength after successful total knee replacement: a 6- to 13-year followup. Clin Orthop Relat Res. 1996 Jul;(328):147-54. doi: 10.1097/00003086-199607000-00023. PMID 8653948
- [Background] Rantanen T, Guralnik JM, Izmirlian G, Williamson JD, Simonsick EM, Ferrucci L, Fried LP. Association of muscle strength with maximum walking speed in disabled older women. Am J Phys Med Rehabil. 1998 Jul-Aug;77(4):299-305. doi: 10.1097/00002060-199807000-00008. PMID 9715919
- [Background] Skelton DA, Greig CA, Davies JM, Young A. Strength, power and related functional ability of healthy people aged 65-89 years. Age Ageing. 1994 Sep;23(5):371-7. doi: 10.1093/ageing/23.5.371. PMID 7825481
- [Background] Moreland JD, Richardson JA, Goldsmith CH, Clase CM. Muscle weakness and falls in older adults: a systematic review and meta-analysis. J Am Geriatr Soc. 2004 Jul;52(7):1121-9. doi: 10.1111/j.1532-5415.2004.52310.x. PMID 15209650
- [Background] Brown M, Sinacore DR, Host HH. The relationship of strength to function in the older adult. J Gerontol A Biol Sci Med Sci. 1995 Nov;50 Spec No:55-9. doi: 10.1093/gerona/50a.special_issue.55. PMID 7493219
- [Background] Connelly DM, Vandervoort AA. Effects of detraining on knee extensor strength and functional mobility in a group of elderly women. J Orthop Sports Phys Ther. 1997 Dec;26(6):340-6. doi: 10.2519/jospt.1997.26.6.340. PMID 9402571
- [Background] Moxley Scarborough D, Krebs DE, Harris BA. Quadriceps muscle strength and dynamic stability in elderly persons. Gait Posture. 1999 Sep;10(1):10-20. doi: 10.1016/s0966-6362(99)00018-1. PMID 10469937
- [Background] LaStayo PC, Meier W, Marcus RL, Mizner R, Dibble L, Peters C. Reversing muscle and mobility deficits 1 to 4 years after TKA: a pilot study. Clin Orthop Relat Res. 2009 Jun;467(6):1493-500. doi: 10.1007/s11999-009-0801-2. Epub 2009 Mar 31. PMID 19333672
- [Background] Meier W, Mizner RL, Marcus RL, Dibble LE, Peters C, Lastayo PC. Total knee arthroplasty: muscle impairments, functional limitations, and recommended rehabilitation approaches. J Orthop Sports Phys Ther. 2008 May;38(5):246-56. doi: 10.2519/jospt.2008.2715. Epub 2007 Dec 14. PMID 18448878
- [Background] Mizner RL, Stevens JE, Snyder-Mackler L. Voluntary activation and decreased force production of the quadriceps femoris muscle after total knee arthroplasty. Phys Ther. 2003 Apr;83(4):359-65. PMID 12665406
- [Background] Rice DA, McNair PJ. Quadriceps arthrogenic muscle inhibition: neural mechanisms and treatment perspectives. Semin Arthritis Rheum. 2010 Dec;40(3):250-66. doi: 10.1016/j.semarthrit.2009.10.001. Epub 2009 Dec 2. PMID 19954822
- [Background] Pichonnaz C, Bassin JP, Lecureux E, Currat D, Jolles BM. Bioimpedance spectroscopy for swelling evaluation following total knee arthroplasty: a validation study. BMC Musculoskelet Disord. 2015 Apr 25;16:100. doi: 10.1186/s12891-015-0559-5. PMID 25907994
- [Background] Pua YH. The Time Course of Knee Swelling Post Total Knee Arthroplasty and Its Associations with Quadriceps Strength and Gait Speed. J Arthroplasty. 2015 Jul;30(7):1215-9. doi: 10.1016/j.arth.2015.02.010. Epub 2015 Feb 19. PMID 25737387
- [Background] Snyder MA, Sympson AN, Scheuerman CM, Gregg JL, Hussain LR. Efficacy in Deep Vein Thrombosis Prevention With Extended Mechanical Compression Device Therapy and Prophylactic Aspirin Following Total Knee Arthroplasty: A Randomized Control Trial. J Arthroplasty. 2017 May;32(5):1478-1482. doi: 10.1016/j.arth.2016.12.027. Epub 2016 Dec 23. PMID 28159420
- [Background] Pichonnaz C, Bassin JP, Lecureux E, Christe G, Currat D, Aminian K, Jolles BM. Effect of Manual Lymphatic Drainage After Total Knee Arthroplasty: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2016 May;97(5):674-82. doi: 10.1016/j.apmr.2016.01.006. Epub 2016 Jan 30. PMID 26829760
- [Background] Wouthuyzen-Bakker M, Lora-Tamayo J, Senneville E, Scarbourough M, Ferry T, Uckay I, Salles MJ, O'Connell K, Iribarren JA, Vigante D, Trebse R, Arvieux C, Soriano A, Ariza J; Group of Investigators for Streptococcal Prosthetic Joint Infection. Erysipelas or cellulitis with a prosthetic joint in situ. J Bone Jt Infect. 2018 Oct 4;3(4):222-225. doi: 10.7150/jbji.25519. eCollection 2018. PMID 30416947
- [Background] Liu P, Mu X, Zhang Q, Liu Z, Wang W, Guo W. Should compression bandage be performed after total knee arthroplasty? A meta-analysis of randomized controlled trials. J Orthop Surg Res. 2020 Feb 14;15(1):52. doi: 10.1186/s13018-019-1527-9. PMID 32059737